CLINICAL TRIAL: NCT00174889
Title: Efficacy and Safety of Pregnenolone Augmentation in the Management of Schizophrenia Patients: a Randomised Double-Blind Placebo-Controlled Trial
Brief Title: Pregnenolone in the Management of Schizophrenia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sha'ar Menashe Mental Health Center (Other)
Collaborators: Beersheva Mental Health Center (Other Government)
Responsible Party: Michael S Ritsner, Shaar-Menashe MHC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PREG 6/2004
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Pregnenolone; Neurosteroids
MeSH Terms: conditions — Schizophrenia | interventions — Pregnenolone

INTERVENTIONS:
Drug: Pregnenolone

SUMMARY:
Pregnenolone is a "neurosteroid" and possesses intrinsic behavioral and brain effects in animals, affecting the GABA(A) and other receptors. Pregnenolone is serves as the precursor for dehydroepiandrosterone (DHEA) and its sulfate ester (DHEAS). There is evidence of efficacy of DHEA augmentation in schizophrenia, we therefore sought to examine the efficacy of augmentation of antipsychotic treatment of schizophrenia patients with pregnenolone. It is hypothesized that the combined effect of antipsychotic agents and pregnenolone would be beneficial in the treatment of negative,depressive, and cognitive symptoms.

DETAILED DESCRIPTION:
Either pregnenolone (30 mg/d or 200 mg/d), DHEA (400 mg/d)or placebo will be added to regular treatment for 8 weeks. Subjects will be assessed at baseline and after 2, 4, 6 and 8 weeks of treatment. An extensive battery of research instruments will be used for assessment of the following domains of interest: psychopathology, insight, side effects, and cognitive functions. Plasma pregnenolone, DHEA(S), cortisol and other relevant steroids will be assayed at baseline, 2, 4, 6 and 8 weeks of treatment. Efficacy and safety of augmentation of antipsychotic treatment with pregnenolone will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for schizophrenia or schizoaffective disorder
* Ability and willingness to sign informed consent for participation in the study

Exclusion Criteria:

* Evidence of organic brain damage, mental retardation, alcohol or drug abuse
* Prostate nodules or cancer.
* Moderate symptoms of benign prostatic hypertrophy such as hesitancy, urgency, frequent voiding and feeling of incomplete voiding.
* History of ischemic cardiac disease.
* Renal disease.
* Hepatic dysfunction.
* Women with a history of carcinoma of the breast, or any women with a family history of the following: premenopausal breast cancer or bilateral breast cancer in a first degree relative; multiple family members (greater than three relatives) with postmenopausal breast cancer.
* Women with a history of uterine cancer.
* Patients with a known hypersensitivity to androgens.
* Pregnant women.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2005-01; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The computerized Cambridge Neuropsychological Test Automated Battery (CANTAB).
The Positive and Negative Syndrome Scale.
The Scale for the Assessment of Negative Symptoms.
The Calgary Depression Scale for Schizophrenia.
The Hamilton Scale for Anxiety.
Extrapyramidal Symptom Rating Scale.
Barnes Akathisia Scale.
Abnormal Involuntary Movement Scale.

SECONDARY OUTCOMES:
The Scale to assess Unawareness of Mental Disorder (SUMD, Amador, 1999).

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Ritsner, MD, PhD, Principal Investigator — Sha'ar Menashe Mental Health Center
Locations (1):
- Sha'ar Menashe Mental Health, Hadera, Israel

REFERENCES:
- [Background] Ritsner M, Gibel A, Ram E, Maayan R, Weizman A. Alterations in DHEA metabolism in schizophrenia: two-month case-control study. Eur Neuropsychopharmacol. 2006 Feb;16(2):137-46. doi: 10.1016/j.euroneuro.2005.07.007. Epub 2005 Sep 1. PMID 16139994
- [Background] Ritsner M, Gibel A, Maayan R, Ratner Y, Ram E, Biadsy H, Modai I, Weizman A. Cortisol/dehydroepiandrosterone ratio and responses to antipsychotic treatment in schizophrenia. Neuropsychopharmacology. 2005 Oct;30(10):1913-22. doi: 10.1038/sj.npp.1300747. PMID 15870835
- [Derived] Ritsner MS, Gibel A, Shleifer T, Boguslavsky I, Zayed A, Maayan R, Weizman A, Lerner V. Pregnenolone and dehydroepiandrosterone as an adjunctive treatment in schizophrenia and schizoaffective disorder: an 8-week, double-blind, randomized, controlled, 2-center, parallel-group trial. J Clin Psychiatry. 2010 Oct;71(10):1351-62. doi: 10.4088/JCP.09m05031yel. Epub 2010 Jun 15. PMID 20584515